CLINICAL TRIAL: NCT05752539
Title: Clinical Evaluation of Implants Restored With Advanced Lithium Disilicate Screw-retained Crowns
Status: Active, not recruiting | Type: Observational
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Other Study IDs: HUM00226401
Record Dates: First submitted 2023-01-16; First posted 2023-03-02 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Dental Prosthesis Failure; Dental Prosthesis Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CEREC System by Dentsply Sirona — CEREC Tessera blocks achieve exceptional three-way performance through a unique chemistry that incorporates two complementary crystal structures within a glassy zirconia matrix. These two crystals work together to create an unprecedented fusion of strength and beauty in one block while significantly improving overall processing time.

SUMMARY:
This is a prospective observational clinical trial to evaluate the clinical performance of the Cerec Tessera prosthetic assembly on implants restored with chairside CAD/CAM-generated crowns. This investigation is intended as a Post Market Clinical Follow-up study for the product Cerec Tessera and its prosthetic assembly for implants, which will serve as a life-cycle approach to safety, backed up by clinical data and post-market monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years.
* Willing and able to sign and date the informed consent form and HIPAA form.
* Have a single implant that has been successfully osseointegrated and deemed ready for restoration by the surgeon placing the implant.

(A maximum of two single dental implant restorations per subject will be restored.)

* Have a single implant that is acceptable to be restored with a digital workflow using the CEREC system.
* Have a single implant to be restored with a screw retained advanced lithium disilicate crown.
* Have a single implant with at least one adjacent tooth contact and with an occlusal contact.

Exclusion Criteria:

* Not willing to participate in the clinical investigation or not able to understand the content of the clinical investigation.
* Unlikely to be able to comply with clinical investigation procedures according to the Principle Investigator's/Co-investigator's judgement.
* Unable or unwilling to return for recall appointments for a period of 5 years.
* Severe non-compliance to Clinical Investigation Protocol as judged by the PI or Co-investigators.
* Women who self-report that they are possibly pregnant, pregnant, or lactating, as elective dental treatment is not indicated at these times.
* Previous enrollment in the present clinical investigation.
* Involvement in the planning and conduct of the clinical investigation (applies to both Dentsply Sirona personnel and from the clinical investigation site).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients in School of Dentistry clinics that have had at least one dental implant placed and ready for restoration. In addition, all subjects enrolled into the study must fulfill below eligibility criterion.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2028-02-20 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of restoration condition measured through Modified FDI criteria | At the 5 years visit
  Modified FDI criteria is based on the questionnaire "The Modified Clinical Evaluation Criteria for Ceramic Crowns" with consists of questions related to: A. Aesthetic properties and B. Functional properties.

SECONDARY OUTCOMES:
Evaluation of restoration condition measured through Modified FDI criteria | At the 4 weeks visit, 9 months visit, 18 months visit, 30 months visit, and at the 4 years visit.
  Modified FDI criteria is based on the questionnaire "The Modified Clinical Evaluation Criteria for Ceramic Crowns" with consists of questions related to: A. Aesthetic properties and B. Functional properties.
Change in bone health compared to baseline (i.e., restoration visit). | At the baseline and restoration visit, 4 weeks visit, 9 months visit, 18 months visit, 30 months visit, 4 years visit, and at the 5 years visit
  The level of the bone around the dental implant will be qualitatively compared to the radiograph taken at the time the restoration was delivered as well as a Mobility Index.

OTHER OUTCOMES:
Evaluation of soft tissue health through Papilla index | At the 4 weeks visit, 9 months visit, 18 months visit, 30 months visit, 4 years visit, and at the 5 years visit
  Papilla contour measurements of the interproximal papilla measured from a reference line through the highest gingival curvatures or the implant crown restoration on the mesio-buccal and disto-buccal side with the adjacent permanent tooth. Papilla index (Jemt, 1997) with gradings from 0 - 4.
Evaluation of soft tissue health through Gingival index | At the 4 weeks visit, 9 months visit, 18 months visit, 30 months visit, 4 years visit, and at the 5 years visit
  Gingival index (based upon the standard Loe & Silness Index, 1963). Gingival score (visual) for gingival area nearest to the crown margin, score 0 - 3.
Evaluation of soft tissue health through Plaque index | At the 4 weeks visit, 9 months visit, 18 months visit, 30 months visit, 4 years visit, and at the 5 years visit
  Plaque index (based upon the standard Silness & Loe Index, 1964). Plaque score (visual) for facial gingival area nearest to the crown margin, score 0 - 3.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J. Fasbinder, DDS, Principal Investigator — Clinical Professor of Dentistry, Department of Cardiology, Restorative Sciences, and Endodontics
Locations (1):
- Department of Cariology, Restorative Sciences, and Endodontics at School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No